CLINICAL TRIAL: NCT00398528
Title: An fMRI Study of Treatment Optimization Recommendations Comparing Patients Changing Treatment From Glatiramer Acetate 20 mg qd SC (Copaxone®) to IFN-β-1a 30 Mcg qw IM (Avonex®) to Those Changing From to IFN-β-1a 30 Mcg qw IM (Avonex®) to Glatiramer Acetate 20 mg qd SC (Copaxone®) in a Multicenter Study of Patients With Relapsing Remitting Multiple Sclerosis Currently on Disease-Modifying Therapy.
Brief Title: An fMRI Study of Treatment Optimization Comparing Two Disease Modifying Therapies Used to Treat Relapsing Remitting Multiple Sclerosis
Status: Terminated | Type: Observational
Why Stopped: rate of enrollment
Sponsor: Neurognostics (Industry)
Other Study IDs: MSAV1-2006
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-11

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Disease Modifying Therapy
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Glatiramer Acetate; Interferon beta-1a

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Glatiramer acetate, (Copaxone®)
Drug: IFN-β-1a, (Avonex®)

SUMMARY:
Impaired short term memory, attention and concentration lapses, and slower processing of information occur in up to 40-65% of patients with Multiple Sclerosis (MS). The quality of life of individuals with MS is impacted to the degree with which they experience these symptoms.

There are several medications approved by the United States Food and Drug Administration (FDA) to treat MS symptoms and to modify (slow) disease course. Traditional approaches to determining the effectiveness of medications used in treating MS rely on reports of the number of relapses an individual experiences, as well as standard clinical tests, such as the Kurtzke Expanded Disability Status Scale (EDSS).

This research study will look at whether the functional magnetic resonance imaging (fMRI) scan can be used as a tool for measuring changes in the brain associated with treatment in MS patients. Unlike a typical MRI which provides structural information about the brain, the fMRI provides information about brain activity during performance of cognitive or motor tasks.

DETAILED DESCRIPTION:
The development of the immunomodulatory, disease-modifying therapies (DMT) represents a major advance for the treatment of multiple sclerosis (MS). To date, immunomodulatory agents approved for the treatment of MS in the United States include two forms of recombinant interferon-beta (IFN-beta-1a [Avonex, Rebif] and IFN-beta-1b [Betaseron]) and synthetic glatiramer acetate [Copaxone].

These drugs have been shown to favorably alter the natural history of relapsing remitting MS by slowing the progression of disability, reducing relapse rate, and decreasing brain inflammation as measured by MRI. There is evidence that the treatment effects of both IFN-beta and glatiramer acetate are related to their properties in regulating various components of the immune system, in particular, the T cell functions (e.g. proliferation and migratory behavior) and cytokine production.

Though demonstrating clear efficacy on a number of short-term clinical measures, these agents are not cures and most patients with MS continue to experience disease activity in spite of treatment. Over the last ten years, clinicians have become comfortable initiating therapy with DMT. Now, attention is focused on monitoring the results of a chosen therapy and deciding whether or not a patient is responding optimally to treatment. At present, however, clinicians lack criteria for defining optimal response to DMT as well as evidence-based recommendations on how to improve treatment outcomes for individual patients.

Using a recently published model generated by an advisory board from the United States, as a framework, The Canadian Multiple Sclerosis Working Group (CMSWG) developed practical, evidence-based recommendations on how neurologists can assess the status of patients on DMT and decide when it may be necessary to modify treatment in order to optimize outcomes. The CMSWG's recommendations are based on monitoring relapses, neurological progression and MRI activity. These recommendations have yet to be implemented in a prospective, randomized, comparative Phase IV clinical trial.

Traditional measures do not provide critical information about the neural systems that underlie change in behavioral performance. The goal of developing a surrogate biological marker of drug efficacy is to be able to measure the extent to which a drug reaches its intended targeted neural system, and to understand and predict the impact of treatment on existing neuropathology. Ideally, relevant clinical outcome measures should be well correlated with the biomarker.

fMRI is a new tool for noninvasive imaging of human brain function. Without the use of contrast agents, fMRI detects regional MR signal increases that have been hypothesized to reflect decreases in deoxyhemoglobin due to local increases in blood flow/volume during task activation. fMRI has higher spatial and temporal resolution than other existing functional imaging techniques, making it ideal for the study of complex cognitive functions in patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization.
* Age between 18 and 65 years
* Male and female subjects with clinically definite or laboratory-supported definite relapsing-remitting multiple sclerosis
* A minimum disease level according to the McDonald criteria for the definition of MS based on results of an MRI scan; acquired within 1 year (Subjects with other significant abnormal findings will be excluded)
* Receiving consistent therapy with Copaxone® or Avonex® for at least 1 year.
* Expanded Disability Status Score (EDSS) of 0 to ≤ 5.5, inclusive
* Exhibiting low or medium level of concern within 12 months prior to screening based on: relapses, or clinical progression, or MRI progression
* Clinical stability or improving neurological state during the eight weeks before Study Day 0
* Willingness & ability to comply with the protocol for the duration of the study
* Confirmation that a subject capable of having children is not pregnant must be established by a negative urine pregnancy test within 30 days of Screening and a negative urine pregnancy test on Scan Days.

Exclusion Criteria:

* Pregnant or lactating women, or women of childbearing potential not using an acceptable method of contraception
* Progressive forms of MS (Primary progressive, Secondary progressive)
* Exhibiting a high level of concern within 12 months prior to screening based on: relapses, or clinical progression, or MRI progression
* Subjects who have been on DMTs other than Copaxone® or Avonex® for longer than 3 months
* Subjects who have been on Avonex® or Copaxone® for less than 3 months and have exhibited intolerability
* History of hypersensitivity to natural or recombinant interferon beta, human serum albumin, or any other component of the Avonex® formulation (for Avonex® Group A)
* History of hypersensitivity to glatiramer acetate or mannitol, or any other component of the Copaxone® formulation (for Copaxone® Group B)
* Participation in any other studies involving investigational or marketed products, concomitantly or within 30 days prior to screening
* Treatment with oral or systemic corticosteroids or ACTH within 4 weeks of screening or ongoing chronic treatment with systemic corticosteroids.
* Treatment with immunomodulatory or immunosuppressive therapy (including but not limited to cyclophosphamide, cyclosporine, methotrexate, azathiprine,linomide, mitoxantrone, Campath) within the 12 months prior to study day 0
* Prior cytokine or anti-cytokine therapy within 3 months prior to Study Day 0
* Prior use of cladribine or have received total lymphoid irradiation
* Have taken intravenous immunoglobulin or any other investigational drug or taken part in any experimental procedure in the 6 months prior to screening
* Psychiatric disorder that is unstable or would preclude safe participation in the study
* Cognitive impairment which impairs ability to understand or comply with the protocol procedures
* Significant leucopenia (white blood cell count <0.5 times the lower limit of normal)as assessed during the course of routine standard of care
* Elevated liver function tests (ALT, AST, alkaline phosphatase or total bilirubin >2 times the upper limit of normal) as assessed during the course of routine standard of care
* Specific systemic diseases, (including insulin-dependent diabetes, Lyme disease,clinically significant cardiac disease, HIV, HTLV-1, and Hepatitis B or C), or other uncontrolled major medical conditions (depression, seizure disorder) that would interfere with the participant's safety, compliance or evaluation
* Unable and/or unlikely to follow the protocol for any reason
* Alcohol and/or any other drug abuse
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol
* Abnormal baseline clinical findings considered by the investigator to be indicative of conditions that might affect study results
* Impaired renal function, as shown by but not limited to serum creatinine >2.5 mg/dL
* Subjects who cannot take the FDA approved medication for any reason will be excluded
* Corticosteroids allowed at doses between 500 mg and 1000 mg IV (over 3-5 days for relapses) IV for a maximum of three days

In addition, specific exclusion criteria are required for MRI scanning:

* Ferrous objects within the body
* Pregnancy
* Weight inappropriate for height
* Low visual acuity that cannot be corrected with glasses
* History of claustrophobia
* Participants whose high-resolution anatomic MR scans reveal the presence of a structural abnormality (other than MS).
* Standard protocol for monitoring based on FDA approved medication will be followed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2006-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Examine the change in task-activated fMRI response as a function of disease modifying therapies assigned to MS.
Secondary: fMRI as a surrogate marker for drug efficacy

SECONDARY OUTCOMES:
fMRI as a surrogate marker for drug efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine L Elsinger, PhD, Study Director — Neurognostics, Inc.; Stephen M Rao, PhD, Principal Investigator — Neurognostics, Inc.
Locations (5):
- United States (5):
  - University of Southern California, Los Angeles, California
  - Minor & James Medical, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin